CLINICAL TRIAL: NCT00994097
Title: NGR014: Randomized Phase II Study of NGR-hTNF in Combination With Standard Chemotherapy Versus Standard Chemotherapy Alone in Previously Untreated Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: NGR-hTNF in Combination With Standard Chemotherapy to Treat Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NGR014; 2008-002703-20 (EudraCT Number)
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NGR-hTNF; Randomized controlled trial; Gemcitabine; Cisplatin; Pemetrexed; Carcinoma, non-small cell lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human; Cisplatin; Gemcitabine; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: NGR-hTNF + cisplatin/gemcitabine or cisplatin/pemetrexed (Experimental): NGR-hTNF with cisplatin/gemcitabine regimen in patients with squamous histology or with cisplatin/pemetrexed regimen in patients with nonsquamous histology
  Interventions: Drug: NGR-hTNF; Drug: Cisplatin; Drug: Gemcitabine; Drug: Pemetrexed
- B: cisplatin/gemcitabine or cisplatin/pemetrexed (Active Comparator): Cisplatin/gemcitabine regimen is administered in patients with squamous histology and cisplatin/pemetrexed regimen is administered in patients with nonsquamous histology
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Pemetrexed

INTERVENTIONS:
Drug: NGR-hTNF — NGR-hTNF: 0.8 mcg/m² as 60-minute intravenous infusion every 3 weeks until confirmed evidence of disease progression or unacceptable toxicity occurs
  Arms: A: NGR-hTNF + cisplatin/gemcitabine or cisplatin/pemetrexed
Drug: Cisplatin — Cisplatin: 80 mg/m² intravenous infusion on day 1 every 3 weeks for a maximum of 6 cycles
Drug: Gemcitabine — Gemcitabine: 1,250 mg/m² intravenous infusion on days 1 and 8 every 3 weeks for a maximum of 6 cycles
Drug: Pemetrexed — Pemetrexed: 500 mg/m² intravenous infusion on day 1 every 3 weeks for a maximum of 6 cycles

SUMMARY:
The main objective of this study is to demonstrate superiority in progression-free survival (PFS) when NGR-hTNF is added to standard chemotherapy regimen (cisplatin/gemcitabine or cisplatin/pemetrexed) in locally advanced (stage IIIb with supraclavicular lymph node metastases or malignant pleural or pericardial effusion), metastatic (stage IV) or recurrent non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Eligible patients will be randomly assigned to a standard chemotherapy regimen plus low-dose (0.8 mcg/m^2) NGR-hTNF or standard chemotherapy alone, through a centralized randomization process using the following stratification factors: performance status (0 vs 1) and histology (squamous vs non-squamous). In both arms the choice between the two chemotherapy regimens will be based on the histologic subtype: in patients with squamous histology (including also generic diagnosis of NSCLC without further subtype classification) is recommended cisplatin/gemcitabine regimen, in patients with nonsquamous histology (including adenocarcinoma and large-cell carcinoma) is recommended cisplatin/pemetrexed regimen.

ELIGIBILITY:
Inclusion criteria:

1. Histologically or cytologically documented inoperable, locally advanced (stage IIIb with supraclavicular lymph node metastases or malignant pleural or pericardial effusion), metastatic (stage IV) or recurrent NSCLC. Mixed tumors should be categorized according to the predominant cell type.
2. Age ≥18 years
3. Life expectancy more than 3 months
4. ECOG performance status 0-1
5. At least one unidimensional measurable lesion (as per RECIST criteria)
6. Adequate baseline bone marrow, hepatic and renal function, defined as follows:

   * Neutrophils >1.5 x 10^9/L and platelets > 100 x 10^9/L
   * Bilirubin <1.5 x ULN
   * AST and/or ALT <2.5 x ULN in absence of liver metastasis
   * AST and/or ALT <5 x ULN in presence of liver metastasis
   * Serum creatinine <1.5 x ULN
   * Creatinine clearance (estimated according to Cockcroft-Gault formula) ≥ 50 ml/min
7. Patients may have had prior therapy providing the following conditions are met:

   * Radiation therapy: wash-out period of 28 days
   * Surgery: wash-out period of 14 days
8. Patients must give written informed consent to participate in the study

Exclusion criteria:

1. Prior chemotherapy or treatment with another systemic anti-cancer agent (for example monoclonal antibody, tyrosine kinase inhibitor).
2. Patients must not receive any other investigational agents while on study
3. Patients with myocardial infarction within the last six (6) months, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
4. Uncontrolled hypertension
5. Prolonged QTc interval (congenital or acquired)
6. Patient with significant peripheral vascular disease
7. History or evidence upon physical examination of CNS disease unless adequately treated (e.g., primary brain tumor, any brain metastasis, seizure not controlled with standard medical therapy, or history of stroke).
8. Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
9. Known hypersensitivity/allergic reaction or contraindications to human albumin preparations or to any of the excipients
10. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
11. Pregnancy or lactation. Patients - both males and females - with reproductive potential (i.e. menopausal for less than 1-year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of child-bearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Every 6 weeks during study treatment and every 6 weeks during the follow-up before PD
  PFS evaluated according to Response evaluation criteria in solid tumors (RECIST)

SECONDARY OUTCOMES:
Safety according to NCI-CTCAE criteria (version 3) | from the date of randomization until 28 days after last treatment
  To evaluate safety profile related to NGR-hTNF in combination with standard chemotherapy
Objective response rate | Every 6 weeks during study treatment and every 6 weeks during the follow-up before PD
  Antitumor activity defined as response rate evaluated according to Response evaluation criteria in solid tumors (RECIST)
Duration of response (DR) | from the time of first recorded evidence of complete response or partial response until the progressive disease objectively documented
  defined as the time that measurement criteria are met for complete response or partial response (whichever status is recorded first) until the progressive disease is objectively documented.
Overall survival (OS) | from the randomization until to the date of patient death or discontinuation from the study
  Defined as the time from the date of randomization until the date of death due to any cause or the last date the patient was known to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lambiase, MD, Study Director — AGC Biologics S.p.A.
Locations (4):
- Italy (4):
  - Istituto Nazionale per la ricerca sul cancro, Genoa
  - Fondazione San Raffaele del Monte Tabor, Milan
  - Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo Oncologico, Milan